CLINICAL TRIAL: NCT05202613
Title: Non-Interventional Observational Retrospective Study to Evaluate Doravirine Based-regimens in HIV Infected Aged Patients (DORAge).
Acronym: DORAge
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Prof. Gabriella d'Ettorre, Professor, University of Roma La Sapienza
Other Study IDs: 6496
Record Dates: First submitted 2022-01-11; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: HIV
Keywords: HIV; Doravirine; Virological Failure; Metabolism; Inflammation
MeSH Terms: conditions — Inflammation | interventions — doravirine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dorage group: * HIV-1 infected patients
  * aged > 50 years old
  * naive patients receiving doravirine-based regimens
  * experienced patients with persistent HIV RNA < 50 copies/mLfor at least 6 months, who switched to doravirine-based regimens, because of toxicity, convenience or other reasons.
  Interventions: Drug: Doravirine
- Control group: HIV negative subjects, matched for age and Charlson Index score (to evaluate comorbidity impact)

INTERVENTIONS:
Drug: Doravirine — Doravirine, both as single drug and as fixed combination with lamivudine and tenofovir disoproxil fumarate
  Groups: Dorage group

SUMMARY:
The HIV-infected population is aging due to the success of combination antiretroviral therapy, which prolongs survival, as well as the growing number of newly diagnosed cases in adults 50 years old and over. This real-life, observational and retrospective study aims to evaluate the virological efficacy, toxicity and tolerability of Doravirine-based regimens in aged HIV-1 positive patients (> 50 years), focusing on metabolic patterns and inflammation markers.

DETAILED DESCRIPTION:
HIV-infected individuals suffer from an accelerated aging due to the persistent and chronic activation of the immune system that leads to immune exhaustion and accelerated immunosenescence. The success of combination antiretroviral therapy, which also prolongs patients' survival, have relatively higher retention rates among HIV infected elderly patients, but only a small percentage are virally suppressed, largely due to elderly drugs interacts with ART and several comorbidities that reduces the life span of elderly people.

In this context, Doravirine is the only NNRTI with a low propensity for resistance, excellent tolerability, a superior neuropsychiatric profile compared with EFV, a superior lipid profile compared with ritonavir-boosted darunavir and EFV, minimal risk for drug- drug interactions, and no food restrictions. In addition, doravirine has a large therapeutic index and robust efficacy in patients with high viral load. However, to date, data on doravirine in HIV aged patients are still lacking.

This observational retrospective cohort in real world will aim to describe the effect of doravirine regimens, both as single drug and as fixed combination with lamivudine and tenofovir disoproxil fumarate, in aged HIV patients.

* The primary endpoint will be the evaluation of virological efficacy defined as the proportion of patients with HIV RNA < 50 copies/mL at the end of the 48-week follow-up.
* The secondary endpoints will be the following:

  * Change in CD4+, CD8 cell counts, CD4/ CD8 ratio from baseline to 48 weeks
  * Proportion of patients with any adverse events (AE), serious adverse events (SAE), also according to their severity.
  * Changes in total HDL and LDL-cholesterol, triglycerides, creatinine, eGFR, phosphate, AST, ALT, FIB-4, ALP, glucose, proteinuria from baseline to 48 weeks.
  * Changes of infiammatory biomarkers: D-Dimer, hsCRP and IL-6 during 48 weeks
  * Occurrence of genotypic mutations (genotypic test) in plasma samples from patients with virological failure

Clinical data will be collected from medical records and laboratory analyses comprising CD4+ T cell count, plasma HIV-1 RNA, blood cells, and plasma chemistry profiles, including fasting lipids (total cholesterol, high-density lipoprotein cholesterol [HDL], low- density lipoprotein [LDL] cholesterol, triglycerides) will be recorded.

The Time horizon for patient follow-up for outcome is at least 12 months (Baseline, 12, 24, 36, 48 weeks).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected patients
* aged > 50 years old
* naive patients receiving doravirine-based regimens both as single drug and as in fixed combination with lamivudine and tenofovir disoproxil fumarate
* experienced patients with persistently undetectable plasma HIV viral load (HIV RNA < 50 copies/mL) for at least 6 months, who switched from any antiretroviral drug to doravirine-based regimens, both as single drug and as fixed combination with lamivudine and tenofovir disoproxil fumarate, because of toxicity, convenience or other reasons.
* estimated creatinine clearance (CrCl) ≥50mL/min.

Exclusion Criteria:

* previous genotypic testing showing resistance mutations to doravirine
* acute hepatitis, decompensated liver disease, liver cirrhosis
* use of systemic immunosuppressive therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV infected patients
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Virological efficacy | 48 weeks
  Assessing the virological efficacy (HIV RNA < 50 copies/mL) of the Doravirine regimen at the end of the follow-up.

SECONDARY OUTCOMES:
Time to virological failure | 48 weeks
Immunological changes | Baseline to 48 weeks
  Change in CD4+, CD8 cell counts, CD4/ CD8 ratio
Safety profile | Baseline to 48 weeks
  Proportion of patients with any adverse events (AE), serious adverse events (SAE), also according to their severity.
Lipid and metabolic profile | Baseline to 48 weeks
  Changes in total HDL and LDL-cholesterol, triglycerides, creatinine, eGFR, phosphate, AST, ALT, FIB-4, ALP, glucose, proteinuria
Infiammatory biomarkers | 48 weeks
  Evaluation of D-Dimer, hsCRP and IL-6
Resistance profile in patients with virological rebound | Baseline to 48 weeks
  Evaluation of of genotypic mutations occurrence (genotypic test) in plasma samples from patients with virological failure

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Public Health and Infectious Diseases, Rome, Italy/RM, Italy